CLINICAL TRIAL: NCT02727309
Title: A Pilot Study of Second-line Treatment With Apatinib After Trans Arterial Chemoembolization (TACE) in Advanced Hepatocellular Carcinoma Patients
Brief Title: A Study of Second-line Treatment With Apatinib After TACE in Advanced Hepatocellular Carcinoma Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhuxu, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBH001
Record Dates: First submitted 2016-03-28; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Apatinib; Second-line Treatment; Hepatocellular Cancer; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — apatinib

ARMS (1):
- apatinib (Experimental): Patients with advanced hepatocellular carcinoma after been treated with TACE receive apatinib (750mg) daily, until disease progression or unacceptable toxicity.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib: 750 mg is administered orally daily, until disease progression or untolerable toxicity.

SUMMARY:
This study is designed to evaluate the efficacy and safety of TACE combined with apatinib in treating advanced hepatocellular carcinoma. The primary endpoint is progression-free survival (PFS), 3-month PFS, 6-month PFS and 1-year PFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic or cytologic diagnosis of hepatocellular carcinoma
* Have progressed after systematic chemotherapy/target therapy, or cannot tolerated with first-line treatment
* The previous chemotherapy and the present trial registration must be at least 2 weeks apart. And they must have recovered from any toxicity of a previous chemotherapy
* Patients with Child Pugh Class A & B disease are eligible for the study
* Patients with Barcelona Clinic Liver Cancer stage B or C are eligible for the study
* Eastern Cooperative Oncology Group performance score (PS): 0-2
* Life expectancy of at least 12 weeks
* Hepatitis B virus DNA<2000 IU/ml
* Adequate organ function meeting the following:

  * Bone marrow: absolute neutrophil count ≥1.5×109/L (1500/mm3); platelet ≥ 75×109/L; hemoglobin ≥9 g/dL
  * Liver: Serum bilirubin ≤ 1.5 ×ULN, AST and ALT ≤ 5 ×ULN, ALB ≥ 29 g/L
  * Kidney: Cr ≤1.5 ×upper limit of normal
* Within 7 days prior to the start of therapy, women of child-bearing potential must undergo a pregnancy test, which must be negative; men of child-bearing potential: contraceptive measures must be adopted during treatment and within 8 weeks afterward
* Subjects who understand and voluntarily signed a written informed consent form

Exclusion Criteria:

* Previous locoregional therapy within 4 weeks prior to enrollment
* Diagnosed with cholangiocellular carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma
* Prepared for liver transplantation
* Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction)
* A previous history of Interstitial pulmonary disease, drug-induced interstitial disease, radiation pneumonitis requiring hormonal therapy or active interstitial lung disease with any clinical evidence
* Use of CYP3A4 inhibitor within 7 days or CYP3A4 inducer within 12 days prior to enrollment
* Patients with central nervous system metastases or brain metastasis
* Previous definite diagnosis of neuropsychiatric disturbances, including epilepsy or dementia
* Pregnant or lactating women
* Patients with bone metastasis received palliative radiation within 4 weeks prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months
  A duration from the date of initial treatment with apatinib to disease progression(as defined by RECIST) or death.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival (OS) was calculated from the date of initial treatment with apatinib to the date of death due to any cause
Objective response rates | 1.5 months
  Number of participants who achieve complete response or partial response. Either complete response (CR) or partial response (PR) will be evaluated by RECIST, confirmed at least 6 weeks following the date of the initial response.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Department of Interventional Therapy, Beijing, Beijing Municipality, China